CLINICAL TRIAL: NCT07357116
Title: Alteration of the Risk of CArdiovascular DIseases After Pneumonia: a Nationwide Observational Study Using the French Healthcare Claim Database
Brief Title: Alteration of the Risk of CArdiovascular DIseases After Pneumonia
Acronym: ARCADIA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0112_1
Record Dates: First submitted 2025-12-03; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia; Cardiovascular Disease (CKD)
Keywords: pneumonia; cardiovascular sidease; observational study; Routinely Collected Health Data; causality
MeSH Terms: conditions — Pneumonia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Exposure is defined as having reported any kind of pneumonia during the inclusion period. Once a participant has developed pneumonia, he or she belongs to the exposed group throughout the follow-up period.
- Unexposed group: The unexposed group is made up of participants who have not developed pneumonia prior to inclusion and who have been matched to a participant in the exposed group on selected confounders.

SUMMARY:
Pneumonia can be acquired in the community (CAP) or during hospitalization (HAP). It is a leading cause of communicable diseases and the second cause of disability-adjusted life-years in the world (Roquilly et al., Shankar-Hari et al.). HAP is a common infectious disease, affecting up to 40% of patients on mechanical ventilation. It is a major global concern, with 500,000 cases treated annually in Europe. Despite European guidelines, the incidence remains high (Roquilly et al.), leading to significant medical consequences. Thanks to improved early detection and appropriate medical management, pneumonia-related mortality has steadily declined over the past decades. As a result, the number of patients surviving with potential long-term sequelae has increased, with risks of pulmonary function abnormalities, psychological disorders, and impaired quality of life (Shankar-Hari et al., Sipilä et al., Corrales-Medina et al., Ahmed et al.).

Cardiovascular and respiratory diseases (CVRD) are the most common pre-existing conditions in patients with pneumonia, with up to 40% of patients presenting these comorbidities at the time of pneumonia diagnosis (Roquilly et al., Nojiri et al.). The risk of severe cardiovascular and respiratory events increases after pneumonia recovery, with 14% of patients developing a CVRD event within the first year post-infection (Corrales-Medina et al., Herridge et al.), representing a 40% relative increase in CVRD risk compared to patients with CVRD without infection (Lai et al., Angriman et al.).

The objective of the ARCADIA study is to describe the incidence of cardiovascular diseases (CVD) in individuals surviving pneumonia and to compare it to that of patients with similar predisposing comorbidities for CVD but without a history of pneumonia. The investigators hypothesize that pneumonia is a cause of CVD so that patients with a history of pneumonia have a higher risk of developing CVD.

DETAILED DESCRIPTION:
Pneumonia is a leading cause of communicable diseases and the second cause of disability-adjusted life-years in the world (Roquilly et al., Shankar-Hari et al.). Pneumonia can be acquired in the community (community-acquired pneumonia, CAP) or during hospitalization (nosocomial, or Hospital-acquired pneumonia, HAP). CAP is classically induced by virulent bacteria (such as Streptococcus pneumoniae) or viruses (Flu), and new pathogenic viruses such as SARS-CoV2 (COVID-19) can rapidly diffuse in the population.

HAP is a common infectious disease, affecting up to 40% of patients on mechanical ventilation. It is a major global concern, with 500,000 cases treated annually in Europe. Despite European guidelines, the incidence remains high (Roquilly et al.), leading to significant medical consequences. Thanks to improved early detection and appropriate medical management, pneumonia-related mortality has steadily declined over the past decades. As a result, the number of patients surviving with potential long-term sequelae has increased, with risks of pulmonary function abnormalities, psychological disorders, and impaired quality of life (Shankar-Hari et al., Sipilä et al., Corrales-Medina et al., Ahmed et al.).

Cardiovascular and respiratory diseases (CVRD) are the most common pre-existing conditions in patients with pneumonia, with up to 40% of patients presenting these comorbidities at the time of pneumonia diagnosis (Roquilly et al., Nojiri et al.). The risk of severe cardiovascular and respiratory events increases after pneumonia recovery, with 14% of patients developing a CVRD event within the first year post-infection (Corrales-Medina et al., Herridge et al.), representing a 40% relative increase in CVRD risk compared to patients with CVRD without infection (Lai et al., Angriman et al.).

The ARCADIA study is part of the HOMI-LUNG project, funded by the Horizon Europe program. HOMI-LUNG is an international and interdisciplinary initiative aiming to better understand the causal links between respiratory infections (such as pneumonia) and the progression of CVRD. Specifically, the project seeks to quantify the burden of CVRD following pneumonia, assess patient acceptability of long-term health alterations, and define pneumonia endotypes with distinct pathobiological mechanisms associated with CVRD exacerbation.

The objective of the ARCADIA study is to describe the incidence of cardiovascular diseases (CVD) in individuals surviving pneumonia and to compare it to that of patients with similar predisposing comorbidities for CVD but without a history of pneumonia. The investigators hypothesize that pneumonia is a cause of CVD so that patients with a history of pneumonia have a higher risk of developing CVD.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age in the month of the index date.
* Exposed group: participants who declared pneumonia between January 1, 2015 and November 30, 2024.
* Unexposed group: participants who did not declare pneumonia between January 1, 2015 and index date and being selected after matching on age, sex, CVD history, chronic kidney disease, diabetes, antihypertensive deliveries, obesity, lipid-lowering treatments, alcohol and tobacco consumption.

Exclusion Criteria:

* Declared pneumonia between January 1, 2012 and December 31, 2014.
* Pneumonia before the age of 18 between January 1, 2015, and the index date.
* Organ transplant receiver for any of the following organs before or within one year after the index date: heart, kidney, lung, liver, and pancreas.
* Identifier that cannot be reliably tracked in the SNDS (such as a fictitious or provisional identifier, or an identifier that, under specific regimen, fails to distinguish same-sex twins in hospital records).
* Death during index hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The French National Health Data System (SNDS) is a database that centralizes health-related data covering over 99% of residents (Tuppin et al.). Its primary objective is to support epidemiological research and health care system evaluation. It enables longitudinal analyses of health care pathways by linking data sources through anonymized identifiers.
  SNDS include information on reimbursed outpatient care and deliveries, hospital discharge summaries and medical procedures, death and related causes and list of pathologies requiring chronic care.
  These datasets collectively enable large-scale population-based studies on health care utilization, costs, morbidity and mortality. SNDS enable epidemiological studies to be conducted with more than 10 years of hindsight on nearly 68 million people.
Sampling Method: Probability Sample
Enrollment: 2000000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
4-points MACE and 5-points MACE | Up to 10 years
  Acute events relating to the following pathologies are the main outcomes of the ARCADIA study:
  * Acute Coronary Syndrome (MeSH Unique ID: D054058)
  * Lower limb revascularization or major amputation
  * Ischemic Stroke (D000083242)
  * Heart Failure (D006333) requiring Hospitalization (D006760) The primary outcome is therefore a composite outcome, called "4-points MACE", defined by the occurrence of at least one acute event related to the previously cited pathologies. The incidence of 4-point MACE will be compared between groups using an incidence density ratio (IDR) and its 95% confidence interval.
  This primary analysis will be replicated by adding all-cause mortality (MeSH Unique ID: D003643) to the 4-point MACE described above, defining a 5-points MACE.

SECONDARY OUTCOMES:
4-points chronic CVD | Up to 10 years
  Secondary outcomes gather chronic CVD as follows:
  * Coronary Artery Disease (MeSH Unique ID: D003324)
  * Peripheral Arterial Disease (D058729)
  * Arterial cerebral disease, non-hemorrhagic
  * Heart failure (D006333) We will also consider a composite outcome, called "4-points chronic cardiovascular disease" (4-points chronic CVD), defined by the occurrence or diagnosis related to these pathologies. Its incidence will be compared between groups using an incidence density ratio (IDR) and its 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ROQUILLY, MD, PhD, Principal Investigator — Nantes Hospital

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Tuppin P, Rudant J, Constantinou P, Gastaldi-Menager C, Rachas A, de Roquefeuil L, Maura G, Caillol H, Tajahmady A, Coste J, Gissot C, Weill A, Fagot-Campagna A. Value of a national administrative database to guide public decisions: From the systeme national d'information interregimes de l'Assurance Maladie (SNIIRAM) to the systeme national des donnees de sante (SNDS) in France. Rev Epidemiol Sante Publique. 2017 Oct;65 Suppl 4:S149-S167. doi: 10.1016/j.respe.2017.05.004. Epub 2017 Jul 27. PMID 28756037
- [Result] Angriman F, Rosella LC, Lawler PR, Ko DT, Wunsch H, Scales DC. Sepsis hospitalization and risk of subsequent cardiovascular events in adults: a population-based matched cohort study. Intensive Care Med. 2022 Apr;48(4):448-457. doi: 10.1007/s00134-022-06634-z. Epub 2022 Feb 10. PMID 35142896
- [Result] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Result] Ahmed H, Patel K, Greenwood DC, Halpin S, Lewthwaite P, Salawu A, Eyre L, Breen A, O'Connor R, Jones A, Sivan M. Long-term clinical outcomes in survivors of severe acute respiratory syndrome and Middle East respiratory syndrome coronavirus outbreaks after hospitalisation or ICU admission: A systematic review and meta-analysis. J Rehabil Med. 2020 May 31;52(5):jrm00063. doi: 10.2340/16501977-2694. PMID 32449782
- [Result] Corrales-Medina VF, Taljaard M, Yende S, Kronmal R, Dwivedi G, Newman AB, Elkind MS, Lyles MF, Chirinos JA. Intermediate and long-term risk of new-onset heart failure after hospitalization for pneumonia in elderly adults. Am Heart J. 2015 Aug;170(2):306-12. doi: 10.1016/j.ahj.2015.04.028. Epub 2015 May 2. PMID 26299228
- [Result] Lai CC, Lee MG, Lee WC, Chao CC, Hsu TC, Lee SH, Lee CC; National Taiwan University Hospital Health Data Science Research Group. Susceptible period for cardiovascular complications in patients recovering from sepsis. CMAJ. 2018 Sep 10;190(36):E1062-E1069. doi: 10.1503/cmaj.171284. PMID 30201613
- [Result] Nojiri S, Itoh H, Kasai T, Fujibayashi K, Saito T, Hiratsuka Y, Okuzawa A, Naito T, Yokoyama K, Daida H. Comorbidity status in hospitalized elderly in Japan: Analysis from National Database of Health Insurance Claims and Specific Health Checkups. Sci Rep. 2019 Dec 27;9(1):20237. doi: 10.1038/s41598-019-56534-4. PMID 31882961
- [Result] Sipila PN, Heikkila N, Lindbohm JV, Hakulinen C, Vahtera J, Elovainio M, Suominen S, Vaananen A, Koskinen A, Nyberg ST, Pentti J, Strandberg TE, Kivimaki M. Hospital-treated infectious diseases and the risk of dementia: a large, multicohort, observational study with a replication cohort. Lancet Infect Dis. 2021 Nov;21(11):1557-1567. doi: 10.1016/S1473-3099(21)00144-4. Epub 2021 Jun 21. PMID 34166620
- [Result] Shankar-Hari M, Ambler M, Mahalingasivam V, Jones A, Rowan K, Rubenfeld GD. Evidence for a causal link between sepsis and long-term mortality: a systematic review of epidemiologic studies. Crit Care. 2016 Apr 13;20:101. doi: 10.1186/s13054-016-1276-7. PMID 27075205
- [Result] Roquilly A, Chanques G, Lasocki S, Foucrier A, Fermier B, De Courson H, Carrie C, Danguy des Deserts M, Gakuba C, Constantin JM, Lagarde K, Holleville M, Blidi S, Sossou A, Cailliez P, Monard C, Oudotte A, Mathieu C, Bourenne J, Isetta C, Perrigault PF, Lakhal K, Rouhani A, Asehnoune K, Guerci P, Tran Dinh A, Chousterman B, Cupaciu A, Dahyot-Fizelier C, Bellier R, Au Duong J, Mansour A, Morel J, Beauplet G, Vibet MA, Feuillet F, Sebille V, Leone M. Implementation of French Recommendations for the Prevention and the Treatment of Hospital-acquired Pneumonia: A Cluster-randomized Trial. Clin Infect Dis. 2021 Oct 5;73(7):e1601-e1610. doi: 10.1093/cid/ciaa1441. PMID 32970811